CLINICAL TRIAL: NCT02654639
Title: An Open-Label, Multi-center, Phase 2 Study of Switch Maintenance With TAS-102 Plus Bevacizumab Following Oxaliplatin or Irinotecan-Based Fluoropyrimidine-Containing Induction Chemotherapy in Patients With Metastatic Colorectal Cancer
Brief Title: Ph 2 Study of TAS-102 / Bevacizumab Maintenance Therapy Post Induction Chemotherapy in Metastatic Colorectal Cancer
Acronym: ALEXANDRIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator left the institution
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0959
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Advanced Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TAS-102 and Bevacizumab (Experimental): Oral TAS-102 and intravenous Bevacizumab.
  Interventions: Drug: TAS-102; Drug: Bevacizumab

INTERVENTIONS:
Drug: TAS-102 — TAS-102 Twice a day by mouth day 1-5 and 8-12
  Other Names: Lonsurf; Avastin
Drug: Bevacizumab — Bevacizumab by intravenous infusion once every 14 days

SUMMARY:
Phase II study of TAS-102 plus bevacizumab switch maintenance therapy in patients with mCRC

DETAILED DESCRIPTION:
Study Drug:

TAS-102 (trifluridine and tipiracil hydrocholoride) and bevacizumab

Dosing Details:

Starting dose of TAS-102 is 35 mg/m2 administered orally twice daily, after meals, for 5 days a week with 2 days rest for 14 days, followed by 14 days rest (1 treatment cycle).

Bevacizumab 5 mg/kg intravenously every 14 days. The treatment cycle repeats every 28 days. Patients may take TAS-102 plus bevacizumab until they exhibit progression of disease, withdraw consent, or experience unacceptable toxicity.This is a single arm study. All patients receive the same study treatment.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Histologically proven, unresectable, evaluable metastatic colorectal cancer
* 16 to 20 weeks of first-line therapy with oxaliplatin, and/or irinotecan-based flourorpyrimidine-containing chemotherapy plus Bevacizumab
* Patients must have stable disease (or better) during the initial induction chemotherapy with first-line chemotherapy.
* No progressive disease at the time of initiation of maintenance therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Adequate organ and marrow function
* Women of child-bearing potential and men must agree to avoid pregnancy
* Patient must start maintenance therapy at least 14 days after the last administered induction chemotherapy but no later than 30 days.

Exclusion Criteria

* Patients whose tumors have progressed on first-line treatment
* Patients with active concurrent malignancy, other than superficial, non-invasive squamous cell carcinoma of the skin or uterine cervix, within the past three years.
* Women who are pregnant or lactating
* Unstable heart disease
* Uncontrolled active infection requiring antibiotics within one week prior to first dose.
* Patients with active CNS malignancy.
* Persistent protein in the urine
* Patients with bowel obstruction or uncontrolled vomiting.
* Patients with serious psychiatric or medical conditions that could interfere with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Salem, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Weinberg BA, Hartley ML, Salem ME. Precision Medicine in Metastatic Colorectal Cancer: Relevant Carcinogenic Pathways and Targets-PART 2: Approaches Beyond First-Line Therapy, and Novel Biologic Agents Under Investigation. Oncology (Williston Park). 2017 Jul 15;31(7):573-80. PMID 28712102

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAS-102 and Bevacizumab
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAS-102 and Bevacizumab
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Length of Progression-Free Survival
Description: Disease progression will be assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI.
Time Frame: From the first occurrence of progression or death, whichever occurred first, assessed up to 2 years.
Population: The study was terminated early due to recruitment difficulties. 4 subjects were enrolled but no outcomes data was collected and no analysis was performed.
Arm/Group | TAS-102 and Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from the time they signed the informed consent until study completion. The period of collection depended on the length of the treatment period. Across all subjects enrolled, this amounted to 8.75 months of AE collection on average.
Arm/Group | TAS-102 and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 and Bevacizumab (N=4)
Neutropenia (Immune system disorders) | 1 (2)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 and Bevacizumab (N=4)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Immune system disorders) | 2 (4)
Pain (General disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
White blood cell decreased (Immune system disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT02654639/Prot_SAP_000.pdf